CLINICAL TRIAL: NCT00306566
Title: A Phase IIa Study to Evaluate Safety, Tolerability, and Immunogenicity of a Melan-A VLP Vaccine in HLA-A2 Positive Patients With Stage II Malignant Melanoma
Brief Title: Safety and Immunogenicity of a Melan-A VLP Vaccine in Early Stage Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CYT004-MelQbG10 02
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: CYT004-MelQbG10

SUMMARY:
The purpose of this study is to monitor a specific cellular immune response in melanoma patients at an early stage of the disease, that have been vaccinated with a Melan-A VLP vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Able and willing to complete all protocol requirements
* Age: 18 years and older
* Histological confirmed stage II melanoma
* HLA-A*0201 haplotype
* Expected survival of at least 6 months
* ECOG performance status of 0 or 1
* Full recovery from surgery
* Adequate organ and bone marrow functions
* Sexually active males should use adequate contraception throughout the study period and 3 months thereafter.
* Females of child bearing potential should use adequate contraception throughout the study period and 3 months thereafter, that can be oral contraception or a double-barrier local contraception (intra-uterine device plus condom or spermicidal gel plus condom), and have a negative serum pregnancy test within 4 weeks prior to the first dose of the vaccine.

Exclusion Criteria:

* Pregnant or nursing
* Use of an investigational drug within 30 days before enrolment
* Active malignancy in the 5 years prior to enrollment other than melanoma, basal cell carcinoma or cervical carcinoma in situ.
* Major surgery within 4 weeks prior to enrollment.
* Current use of an immunosuppressive drug or any concomitant medication that could potentially interfere with the study drug (e.g. steroids, antihistamine drugs; topical or inhalational steroids are permitted).
* Presence of significant cardiovascular, renal, pulmonary, endocrine, infectious, or neurological disorders.
* Serum tests positive for HIV, HBV, HCV.
* Active autoimmune diseases or severe allergies.
* Current diagnosis or history of relevant and severe psychiatric disorder that compromises the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol or to complete the study.
* Blood donation or loss of > 500mL within 8 weeks prior to inclusion.
* Abuse of alcohol or other recreational drugs.
* Previous vaccination with a Melan-A analog peptide.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Lienard, MD, Principal Investigator — Centre Pluridisciplinaire d'Oncologie & LICR, CHUV
Locations (1):
- Centre Pluridisciplinaire d'Oncologie & LICR, CHUV, Lausanne, Vaude, Switzerland